CLINICAL TRIAL: NCT03796676
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTI-CENTER STUDY INVESTIGATING THE EFFICACY AND SAFETY OF PF-04965842 CO-ADMINISTERED WITH BACKGROUND MEDICATED TOPICAL THERAPY IN ADOLESCENT PARTICIPANTS 12 TO <18 YEARS OF AGE WITH MODERATE-TO-SEVERE ATOPIC DERMATITIS
Brief Title: JAK1 Inhibitor With Medicated Topical Therapy in Adolescents With Atopic Dermatitis
Acronym: JADE TEEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7451036; JADE TEEN (Other: Alias Study Number); 2018-003804-37 (EudraCT Number)
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis, JAK1 inhibitor
MeSH Terms: conditions — Dermatitis, Atopic | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PF-04965842 100 mg QD (Experimental): active
  Interventions: Drug: PF-04965842
- PF-04965842 200 mg QD (Experimental): active
  Interventions: Drug: PF04965842

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PF-04965842 — 100 mg QD
  Arms: PF-04965842 100 mg QD
Drug: PF04965842 — 200 mg QD
  Arms: PF-04965842 200 mg QD

SUMMARY:
This is a randomized, double blind, placebo controlled, parallel group, Phase 3 study to evaluate the efficacy and safety of PF 04965842 in adolescent participants 12 to <18 years of age with moderate to severe AD.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, parallel group, Phase 3 study to evaluate the efficacy and safety of PF 04965842 in adolescent participants 12 to <18 years of age with moderate to severe AD. Participants will be screened within 28 days prior to the first dose of study intervention to confirm study eligibility. Subjects must have moderate-severe AD involving at least 10% Body Surface Area (BSA); an Investigator Global Assessment (IGA) score of at least 3; an Eczema Area Severity Index (EASI) of at least 16 and Peak Pruritus Numerical Rating Score (NRS) of at least 4 on baseline/Day 1. Eligible subjects will be randomized at the Baseline/Day 1 visit. Approximately 225 participants will be randomized in a 1:1:1 ratio to receive once daily PF 04965842 at 200 mg, 100 mg, or placebo for 12 weeks. Randomization will be stratified by baseline disease severity (moderate [IGA = 3] vs. severe [IGA = 4] AD). The investigational products will be administered QD for 12 weeks. Background therapy (medicated and non-medicated topical therapy) must be applied BID for the duration of the treatment period. The co-primary efficacy endpoints are an IGA score of clear (0) or almost clear (1) with a reduction from baseline of greater than 2 points at Week 12 AND an at least 75% improvement of the EASI score (EASI-75) at week 12. Safety and efficacy assessments will be conducted at the investigator site by a clinical assessor blinded to treatment assignment. Scheduled clinic or telephone study visits for all subjects will occur at Screening, Baseline/Day 1, Day 8 (by phone), Day 15, Day 29, Day 43 (by phone), Day 57, Day 85 (End of treatment/Early termination), Day 113 (End of Study). Participants discontinuing early from the study will undergo a 4 week follow up period.

This study includes an immunogenicity sub study integrated into the last 4 weeks of the main study treatment period. At Week 8, up to approximately 90 participants (up to approximately 30 in each treatment arm) who have completed 8 weeks of treatment with study intervention will receive a tetanus, diphtheria and acellular pertussis combination vaccine (Tdap), and collection of blood samples for the evaluation of immunogenicity at Weeks 8 and 12. Participants of this sub study will complete all other protocol specified procedures in the main study.

At the end of the 12 week study treatment, qualified participants completing the study will have the option to enter the long term extension (LTE) study B7451015.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and to 17 with a minimum body weight of 40 kg
* Diagnosis of atopic dermatitis (AD) for at least 1 year and current status of moderate to severe disease (>= the following scores: BSA 10%, IGA 3, EASI 16, Pruritus NRS severity 4)

Exclusion Criteria:

* Acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation
* Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study
* Prior treatment with JAK inhibitors
* Other active non-AD inflammatory skin diseases or conditions affecting skin
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, malignancies, current or history of certain infections, lymphoproliferative disorders and other medical conditions at the discretion of the investigator
* Pregnant or breastfeeding women, or women of childbearing potential who are unwilling to use contraception

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 287 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (135):
- United States (51):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Madera Family Medical Group, Madera, California
  - Allergy & Asthma Associates of Southern California dba Southern California Research, Mission Viejo, California
  - UC Davis, Sacramento, California
  - Moonshine Research Center, Inc., Doral, Florida
  - Homestead Research Institute, Homestead, Florida
  - Olympian Clinical Research, Largo, Florida
  - Clinical Trials Solutions, Miami, Florida
  - Global Health Clinical Trials Corp, Miami, Florida
  - La Salud Research Clinic, Inc., Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - South Miami Medical & Research Group, Inc., Miami, Florida
  - Ciocca Dermatology, PA, Miami, Florida
  - INTERMED Medical Research Center, Inc, Miami, Florida
  - Suncoast Research Associates, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Pediatric Dermatology Orlando, Orlando, Florida
  - AdventHealth Orlando - Investigational Drug Services, Orlando, Florida
  - Outpatient Service Center-AdventHealth Orlando, Orlando, Florida
  - Pediatric Outpatient Procedures and Sedation, Orlando, Florida
  - NeuroSkeletal Imaging, Orlando, Florida
  - Accel Research Sites - Pure Skin Dermatology & Aesthetics, Orlando, Florida
  - Accel Research Sites - Nona Pediatric Center, Orlando, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Midwest Allergy Sinus Asthma, SC, Normal, Illinois
  - NorthShore University HealthSystem Dermatology Clinical Trials Unit, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Forefront Dermatology S.C., Louisville, Kentucky
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - DermAssociates, LLC, Rockville, Maryland
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Clarkston Skin Research, Clarkston, Michigan
  - Wayne State University / Integrative Biosciences Center, Detroit, Michigan
  - Center for Outpatient Health, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Clinical Research Consortium, Las Vegas, Nevada
  - DermResearch Center of New York, Inc., Stony Brook, New York
  - Synexus Clinical Research US, Inc., Cincinnati, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Synexus Clinical Research US, Inc., Greer, South Carolina
  - Austin Institute for Clinical Research, Inc., Austin, Texas
  - Center for Clinical Studies, LTD.LLP, Webster, Texas
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - West Virginia Research Institute, Morgantown, West Virginia
  - Children's Hospital of Wisconsin Investigational Drug Service, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin Translational Research Unit, Milwaukee, Wisconsin
- Australia (5):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - The Skin Hospital, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - The Royal Children's Hospital, Parkville, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria (vic)
- China (10):
  - The First Affiliated Hospital of Fujian Medical University, Dermatology Department, Fuzhou, Fujian
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Shandong Provincial Institute of Dermatology and Venereology & Shandong Provincial Hospital for Skin, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine/Dermatology Dept, Hangzhou, Zhejiang
  - Xin Hua Hospital Affiliated to Shanghai Jiaotong University School of Medicine/Dermatology, Shanghai
  - Shanghai Dermatology Hospital, Shanghai
- Czechia (11):
  - Lekarna Na Vaclavskem namesti, Kutná Hora
  - Kozni ambulance Kutna Hora, s.r.o, Kutná Hora
  - Dermamedica S.R.O., Náchod
  - Oblastni nemocnice Nachod, Náchod
  - Lekarna u Stribrneho orla, Náchod
  - Mestska poliklinika Praha, Prague
  - Lekarna Cisarska, Prague
  - Synexus Czech S.R.O., Prague
  - Dermatovenerologicka ambulance, Svitavy
  - Lekarna na Hranicni, Svitavy
  - Nemocnice Svitavy, Svitavy
- Germany (5):
  - Universitaetsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Fachklinik Bad Bentheim Thermalsole- und Schwefelbad Bentheim GmbH, Bad Bentheim
  - Universitaetsklinikum Bonn, Bonn
  - MENSINGDERMA research GmbH, Hamburg
  - Uniklinik Muenster, Münster
- Hungary (6):
  - Clinexpert Kft., Budapest
  - Bugát Pál Kórház, Bőrgyógyászati Szakrendelés, Gyöngyös
  - Trial Pharma Kft., Győr
  - Trial Pharma Kft., Kaposvár
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Gyermek Gasztroenterológia II. emelet, Miskolc
  - Trial Pharma Kft., Püspökladány
- Istituto Clinico Humanitas IRCSS - UOC di Dermatologia, Milan, Italy
- Japan (8):
  - Takagi Dermatological Clinic, Obihiro, Hokkaido
  - Dermatology Shimizu Clinic, Kobe, Hyōgo
  - Noguchi Dermatology Clinic, Kamimashiki-gun, Kumamoto
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Kume Clinic, Sakai, Osaka
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Hoshikuma Dermatology・Allergy Clinic, Fukuoka
  - Matsuda Tomoko Dermatological Clinic, Fukuoka
- Latvia (2):
  - Aesthetic dermatology clinic of Prof. J. Kisis, Riga
  - Outpatient Clinic Of Ventspils, Ventspils
- Mexico (8):
  - Clinical Research Institute Saltillo S.A. de C.V., Saltillo, Coahuila
  - Trials in Medicine S.C., Cuauhtémoc, Mexico City
  - Hospital Infantil de México Federico Gómez, Del. Cuauhtemoc, Mexico City
  - Hospital de Jesus, I.A.P., Del. Cuauhtémoc, Mexico City
  - Unidad de Atención Médica e Investigación en Salud, Mérida, Yucatán
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan, Mérida, Yucatán
  - Servicios Hospitalarios de Mexico S.A. de C.V. (Hospital Ángeles Chihuahua), Chihuahua City
  - Sociedad de Metabolismo y Corazón S.C., Veracruz
- Poland (16):
  - KLIMED Marek Klimkiewicz, Bialystok
  - Clinica Dermatoestetica Prywatny Gabinet Dermatologiczny i Alergologiczny, Bydgoszcz
  - Centrum Medyczne SENSEMED, Chorzów
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Niepubliczny Zaklad Opieki Zdrowotnej Przychodnia Specjalistyczna "A-DERM-SERWIS", Częstochowa
  - Neutrum Lekarze M. Hlebowicz i Partnerzy Spolka Partnerska, Gdansk
  - MULTIKLINIKA Salute Sp. z o.o., Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Centrum medyczne PLEJADY, Krakow
  - Krakowskie Centrum Medyczne, Krakow
  - Dermoklinika-Centrum Medyczne s.c. M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Irmed, Piotrkow Trybunalski
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
- Spain (8):
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital General Universitario de Alicante, Alicante
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Consultas Externas Dermatologia Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
  - Servicio de Radiologia Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (3):
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Paller AS, Eichenfield LF, Irvine AD, Flohr C, Wollenberg A, Barbarot S, Bangert C, Spergel JM, Selfridge A, Biswas P, Fan H, Alderfer J, Watkins M, Koppensteiner H. Integrated Efficacy and Safety Analysis of Abrocitinib in Adolescents With Moderate-to-Severe Atopic Dermatitis. Allergy. 2025 Aug;80(8):2213-2224. doi: 10.1111/all.16512. Epub 2025 Mar 3. PMID 40028832
- [Derived] Armstrong AW, Alexis AF, Blauvelt A, Silverberg JI, Feeney C, Levenberg M, Chan G, Zhang F, Fostvedt L. Predicting Abrocitinib Efficacy at Week 12 Based on Clinical Response at Week 4: A Post Hoc Analysis of Four Randomized Studies in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1849-1861. doi: 10.1007/s13555-024-01183-3. Epub 2024 Jun 19. PMID 38896380
- [Derived] Cork MJ, McMichael A, Teng J, Valdez H, Rojo R, Chan G, Zhang F, Myers DE, DiBonaventura M. Impact of oral abrocitinib on signs, symptoms and quality of life among adolescents with moderate-to-severe atopic dermatitis: an analysis of patient-reported outcomes. J Eur Acad Dermatol Venereol. 2022 Mar;36(3):422-433. doi: 10.1111/jdv.17792. Epub 2021 Dec 4. PMID 34743361
- [Derived] Eichenfield LF, Flohr C, Sidbury R, Siegfried E, Szalai Z, Galus R, Yao Z, Takahashi H, Barbarot S, Feeney C, Zhang F, DiBonaventura M, Rojo R, Valdez H, Chan G. Efficacy and Safety of Abrocitinib in Combination With Topical Therapy in Adolescents With Moderate-to-Severe Atopic Dermatitis: The JADE TEEN Randomized Clinical Trial. JAMA Dermatol. 2021 Oct 1;157(10):1165-1173. doi: 10.1001/jamadermatol.2021.2830. PMID 34406366
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 287 adolescent participants were randomized to the study, and 285 adolescent participants received study treatment, including 96 participants in the placebo group, 95 participants in the abrocitinib 100 mg QD group, and 94 participants in the abrocitinib 200 mg QD group.
Groups:
- Placebo: Participants received two PF-04965842-matching placebo tablets QD
- PF-04965842 100mg QD: Participants received one PF-04965842 100 mg tablet and one matching placebo tablet QD
- PF-04965842 200mg QD: Participants received two PF-04965842 100 mg tablets QD
Period: Overall Study
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Started | 96 | 95 | 94
Completed | 90 | 92 | 91
Not Completed | 6 | 3 | 3
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Participant did not complete Week 16 due to COVID-19 impact | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD | Total
Number analyzed (Participants) | 96 | 95 | 94 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (1.7) | 15.1 (1.8) | 14.7 (1.8) | 14.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 38 | 140
  Male | 44 | 45 | 56 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 26 | 25 | 76
  Not Hispanic or Latino | 65 | 63 | 69 | 197
  Unknown or Not Reported | 6 | 6 | 0 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 56 | 52 | 52 | 160
  Black or African American | 3 | 9 | 5 | 17
  Asian | 32 | 31 | 31 | 94
  American Indian or Alaska Native | 1 | 3 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Multiracial | 1 | 0 | 1 | 2
  Not reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of 'Clear' (0) or 'Almost Clear' (1) and ≥2 Points Improvement From Baseline at Week 12
Description: The IGA of Atopic Dermatitis (AD) was scored on a 5-point scale (0-4), reflecting a global consideration of the erythema, induration and scaling. The overall severity of AD was assessed according to the 5-point scale: 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, and 4=Severe. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline to Week 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number of Participants Analyzed refers to the number of participants evaluable for this time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 94 | 89 | 93
Percentage of participants | 24.5 [15.8 to 33.2] | 41.6 [31.3 to 51.8] | 46.2 [36.1 to 56.4]
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 100mg QD; Test type: Superiority; p = 0.0147, Cochran-Mantel-Haenszel; Estimate of difference = 16.7, 95% CI 2-sided [3.5 to 29.9] — Estimate of the difference in percentages of response at Week 12 was calculated by PF-04965842 100 mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 200mg QD; Test type: Superiority; p = 0.0030, Cochran-Mantel-Haenszel; Estimate of difference = 20.6, 95% CI 2-sided [7.3 to 33.9] — Estimate of the difference in percentages of response at Week 12 was calculated by PF-04965842 200 mg minus placebo

2. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response ≥ 75% Improvement From Baseline at Week 12
Description: The EASI quantifies the severity of AD based on both severity of lesion clinical signs and the percent of body surface area (BSA) affected. The EASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of AD. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 94 | 89 | 93
Percentage of participants | 41.5 [31.5 to 51.4] | 68.5 [58.9 to 78.2] | 72.0 [62.9 to 81.2]
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 100mg QD; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Estimate of difference = 26.5, 95% CI 2-sided [13.1 to 39.8] — Estimate of the difference in percentages of response at Week 12 was calculated by PF-04965842 100 mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 200mg QD; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Estimate of difference = 29.4, 95% CI 2-sided [16.3 to 42.5] — Estimate of the difference in percentages of response at Week 12 was calculated by PF-04965842 200 mg minus placebo

3. Secondary Outcome: Percentage of Participants Achieving ≥4 Points Improvement From Baseline in Peak Pruritis Numeric Rating Scale (PP-NRS) for Severity of Pruritus at Weeks 2, 4 and 12
Description: PP-NRS assesses the severity of itch (pruritus) due to AD. Participants were asked to assess their worst itching due to AD on an NRS anchored by the terms "no itch" (0) and "worst itch imaginable" (10). Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline, Weeks 2, 4 and 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number of Participants Analyzed refers to the number of participants who were evaluable for this outcome measure. Number analyzed refers to the number of participants evaluable for each time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 95 | 92 | 88
Percentage of participants
  Week 2 | 12.6 [6.0 to 19.3] | 27.2 [18.1 to 36.3] | 38.6 [28.5 to 48.8]
  Week 4: number analyzed (Participants) | 92 | 89 | 84
  Week 4 | 20.7 [12.4 to 28.9] | 31.5 [21.8 to 41.1] | 50.0 [39.3 to 60.7]
  Week 12: number analyzed (Participants) | 84 | 76 | 74
  Week 12 | 29.8 [20.0 to 39.5] | 52.6 [41.4 to 63.9] | 55.4 [44.1 to 66.7]
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 100mg QD; Test type: Superiority; p = 0.0119, Cochran-Mantel-Haenszel; Estimate of difference = 14.7, 95% CI [3.5 to 25.9] — Estimate of the difference in percentages of response at Week 2 was calculated by PF-04965842 100 mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 200mg QD; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Estimate of difference = 26.1, 95% CI 2-sided [13.9 to 38.3] — Estimate of the difference in percentages of response at Week 2 was calculated by PF-04965842 200 mg minus placebo
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 100mg QD; Test type: Superiority; p = 0.0971, Cochran-Mantel-Haenszel; Estimate of difference = 10.9, 95% CI 2-sided [-1.8 to 23.6] — Estimate of the difference in percentages of response at Week 4 was calculated by PF-04965842 100 mg minus placebo
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200mg QD; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Estimate of difference = 29.4, 95% CI 2-sided [16.0 to 42.9] — Estimate of the difference in percentages of response at Week 4 was calculated by PF-04965842 200 mg minus placebo
Statistical Analysis 5: Comparison: Placebo vs PF-04965842 100mg QD; Test type: Superiority; p = 0.0035, Cochran-Mantel-Haenszel; Estimate of difference = 22.8, 95% CI 2-sided [8.0 to 37.7] — Estimate of the difference in percentages of response at Week 12 was calculated by PF-04965842 100 mg minus placebo
Statistical Analysis 6: Comparison: Placebo vs PF-04965842 200mg QD; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; Estimate of difference = 25.6, 95% CI 2-sided [10.6 to 40.6] — Estimate of the difference in percentages of response at Week 12 was calculated by PF-04965842 200 mg minus placebo

4. Secondary Outcome: Change From Baseline in Pruritus and Symptoms Assessment for Atopic Dermatitis (PSAAD) at Week 12
Description: The PSAAD is a daily patient reported symptom diary presented as a 15 item questionnaire that includes 11 items developed to measure symptoms of AD, along with 4 additional items for exploratory and psychometric validation purposes (Sleep & Usual Activities Questions and Patient Global Impression of Severity & Patient Global Impression of Change Questions). Participants answer each question about skin condition based on a 24 hour recall. Each question was evaluated on a 11-point scale ranging from 0 to 10, where higher scores indicate more impact on skin condition.The PSAAD total score is calculated as the average of the responses to each of the 11 items and ranges from 0 (none) to 10 (extreme), where higher scores indicate worse severity of AD symptoms.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 95 | 95 | 93
Units on a scale | -2.0 [-2.4 to -1.6] | -2.5 [-2.9 to -2.1] | -2.7 [-3.1 to -2.3]
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 100mg QD; Test type: Superiority; p = 0.0664, Mixed Models Analysis; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.1 to 0.0] — The least squares mean difference at Week 12 was calculated by PF-04965842 100 mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 200mg QD; Test type: Superiority; p = 0.0142, Mixed Models Analysis; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.3 to -0.1] — The least squares mean difference at Week 12 was calculated by PF-04965842 200 mg minus placebo

5. Secondary Outcome: Percentage of Participants Achieving IGA Response of 'Clear' or 'Almost Clear' and ≥2 Points Improvement From Baseline at All Scheduled Time Points Except Week 12
Description: The IGA of AD is scored on a 5-point scale (0-4), reflecting a global consideration of the erythema, induration and scaling. The overall severity of AD was assessed according to the 5-point scale: 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, and 4=Severe. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline, Weeks 2, 4 and 8
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 92 | 94
Percentage of participants
  Week 2: number analyzed (Participants) | 91 | 92 | 94
  Week 2 | 1.1 [0.0 to 3.2] | 6.5 [1.5 to 11.6] | 12.8 [6.0 to 19.5]
  Week 4 | 3.1 [0.0 to 6.6] | 19.6 [11.5 to 27.7] | 38.3 [28.5 to 48.1]
  Week 8: number analyzed (Participants) | 94 | 91 | 92
  Week 8 | 16.0 [8.6 to 23.4] | 30.8 [21.3 to 40.3] | 48.9 [38.7 to 59.1]

6. Secondary Outcome: Percentage of Participants Achieving EASI Response ≥ 75% Improvement From Baseline at All Scheduled Time Points Except Week 12
Description: The EASI quantifies the severity of AD based on both severity of lesion clinical signs and the percent of BSA affected. The EASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of AD. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline, Weeks 2, 4 and 8
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 92 | 94
Percentage of participants
  Week 2: number analyzed (Participants) | 91 | 92 | 94
  Week 2 | 4.4 [0.2 to 8.6] | 19.6 [11.5 to 27.7] | 25.5 [16.7 to 34.3]
  Week 4 | 14.6 [7.5 to 21.6] | 41.3 [31.2 to 51.4] | 63.8 [54.1 to 73.5]
  Week 8: number analyzed (Participants) | 93 | 91 | 92
  Week 8 | 33.3 [23.8 to 42.9] | 60.4 [50.4 to 70.5] | 68.5 [59.0 to 78.0]

7. Secondary Outcome: Percentage of Participants Achieving EASI Response ≥ 50% Improvement From Baseline
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 92 | 94
Percentage of participants
  Week 2: number analyzed (Participants) | 91 | 92 | 94
  Week 2 | 24.2 [15.4 to 33.0] | 55.4 [45.3 to 65.6] | 64.9 [55.2 to 74.5]
  Week 4 | 51.0 [41.0 to 61.0] | 75.0 [66.2 to 83.8] | 81.9 [74.1 to 89.7]
  Week 8: number analyzed (Participants) | 93 | 91 | 92
  Week 8 | 65.6 [55.9 to 75.2] | 85.7 [78.5 to 92.9] | 82.6 [74.9 to 90.4]
  Week 12: number analyzed (Participants) | 94 | 89 | 93
  Week 12 | 69.1 [59.8 to 78.5] | 87.6 [80.8 to 94.5] | 87.1 [80.3 to 93.9]

8. Secondary Outcome: Percentage of Participants Achieving EASI Response ≥ 90% Improvement From Baseline
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 92 | 94
Percentage of participants
  Week 2: number analyzed (Participants) | 91 | 92 | 94
  Week 2 | 0 [0.0 to 4.0] | 8.7 [2.9 to 14.5] | 10.6 [4.4 to 16.9]
  Week 4 | 2.1 [0.0 to 4.9] | 17.4 [9.6 to 25.1] | 30.9 [21.5 to 40.2]
  Week 8: number analyzed (Participants) | 93 | 91 | 92
  Week 8 | 14.0 [6.9 to 21.0] | 29.7 [20.3 to 39.1] | 40.2 [30.2 to 50.2]
  Week 12: number analyzed (Participants) | 94 | 89 | 93
  Week 12 | 18.1 [10.3 to 25.9] | 41.6 [31.3 to 51.8] | 49.5 [39.3 to 59.6]

9. Secondary Outcome: Percentage of Participants Achieving EASI Response =100% Improvement From Baseline
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 92 | 94
Percentage of participants
  Week 2: number analyzed (Participants) | 91 | 92 | 94
  Week 2 | 0 [0.0 to 4.0] | 1.1 [0.0 to 3.2] | 0 [0.0 to 3.8]
  Week 4 | 0 [0.0 to 3.8] | 2.2 [0.0 to 5.2] | 5.3 [0.8 to 9.9]
  Week 8: number analyzed (Participants) | 93 | 91 | 92
  Week 8 | 0 [0.0 to 3.9] | 3.3 [0.0 to 7.0] | 9.8 [3.7 to 15.9]
  Week 12: number analyzed (Participants) | 94 | 89 | 93
  Week 12 | 2.1 [0.0 to 5.0] | 2.2 [0.0 to 5.3] | 8.6 [2.9 to 14.3]

10. Secondary Outcome: Percent Change From Baseline in EASI Score
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 92 | 94
Percent change
  Week 2: number analyzed (Participants) | 91 | 92 | 94
  Week 2 | -27.6 [-34.0 to -21.2] | -51.5 [-57.9 to -45.1] | -54.5 [-61.0 to -48.0]
  Week 4 | -41.7 [-48.3 to -35.1] | -66.1 [-72.7 to -59.4] | -74.3 [-81.0 to -67.5]
  Week 8: number analyzed (Participants) | 93 | 91 | 92
  Week 8 | -57.6 [-63.4 to -51.8] | -72.6 [-78.4 to -66.8] | -77.8 [-83.7 to -71.9]
  Week 12: number analyzed (Participants) | 94 | 89 | 93
  Week 12 | -63.7 [-69.5 to -57.9] | -77.3 [-83.1 to -71.5] | -80.6 [-86.5 to -74.8]

11. Secondary Outcome: Percentage of Participants Achieving ≥4 Points Improvement From Baseline in PP-NRS for Severity of Pruritus at All Scheduled Time Points Other Than Weeks 2, 4 and 12
Description: as for outcome 3
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 84 | 83 | 82
Percentage of participants
  Day 2: number analyzed (Participants) | 81 | 71 | 77
  Day 2 | 1.2 [0.0 to 3.6] | 2.8 [0.0 to 6.7] | 3.9 [0.0 to 8.2]
  Day 3: number analyzed (Participants) | 79 | 79 | 78
  Day 3 | 0 [0.0 to 4.6] | 5.1 [0.2 to 9.9] | 7.7 [1.8 to 13.6]
  Day 4: number analyzed (Participants) | 81 | 78 | 77
  Day 4 | 4.9 [0.2 to 9.7] | 11.5 [4.4 to 18.6] | 14.3 [6.5 to 22.1]
  Day 5: number analyzed (Participants) | 72 | 82 | 81
  Day 5 | 6.9 [1.1 to 12.8] | 12.2 [5.1 to 19.3] | 18.5 [10.1 to 27.0]
  Day 6: number analyzed (Participants) | 80 | 81 | 80
  Day 6 | 8.8 [2.6 to 14.9] | 16.0 [8.1 to 24.0] | 21.3 [12.3 to 30.2]
  Day 7: number analyzed (Participants) | 79 | 81 | 80
  Day 7 | 10.1 [3.5 to 16.8] | 16.0 [8.1 to 24.0] | 21.3 [12.3 to 30.2]
  Day 8: number analyzed (Participants) | 75 | 75 | 76
  Day 8 | 4.0 [0.0 to 8.4] | 17.3 [8.8 to 25.9] | 25.0 [15.3 to 34.7]
  Day 9: number analyzed (Participants) | 83 | 75 | 80
  Day 9 | 6.0 [0.9 to 11.1] | 16.0 [7.7 to 24.3] | 25.0 [15.5 to 34.5]
  Day 10: number analyzed (Participants) | 84 | 77 | 80
  Day 10 | 8.3 [2.4 to 14.2] | 15.6 [7.5 to 23.7] | 28.8 [18.8 to 38.7]
  Day 11: number analyzed (Participants) | 79 | 77 | 74
  Day 11 | 7.6 [1.8 to 13.4] | 20.8 [11.7 to 29.8] | 27.0 [16.9 to 37.1]
  Day 12: number analyzed (Participants) | 74 | 72 | 72
  Day 12 | 10.8 [3.7 to 17.9] | 22.2 [12.6 to 31.8] | 23.6 [13.8 to 33.4]
  Day 13: number analyzed (Participants) | 80 | 80 | 77
  Day 13 | 10.0 [3.4 to 16.6] | 26.3 [16.6 to 35.9] | 31.2 [20.8 to 41.5]
  Day 14: number analyzed (Participants) | 84 | 81 | 74
  Day 14 | 9.5 [3.2 to 15.8] | 24.7 [15.3 to 34.1] | 32.4 [21.8 to 43.1]
  Day 15 | 14.3 [6.8 to 21.8] | 27.7 [18.1 to 37.3] | 37.8 [27.3 to 48.3]

12. Secondary Outcome: Time to First Achieve ≥4 Points Improvement From Baseline in PP-NRS for Severity of Pruritus
Description: PP-NRS assesses the severity of itch (pruritus) due to AD. Participants were asked to assess their worst itching due to AD on an NRS anchored by the terms "no itch" (0) and "worst itch imaginable" (10).
Time Frame: Baseline to Week 16
Population: The Full Analysis Set (FAS) included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants in the FAS with a baseline numeric rating score for severity of pruritus >=4 were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 93 | 90
Days | 90.0 [62.0 to NA] — The upper limit was not evaluable as too few events were observed. | 70.0 [30.0 to 85.0] | 29.0 [15.0 to 61.0]

13. Secondary Outcome: Percent Change From Baseline in PP-NRS for Severity of Pruritus
Description: as for outcome 12
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 84 | 83 | 82
Percent change
  Day 2: number analyzed (Participants) | 81 | 71 | 77
  Day 2 | -0.9 [-5.5 to 3.6] | -9.5 [-14.2 to -4.8] | -5.4 [-10.0 to -0.7]
  Day 3: number analyzed (Participants) | 79 | 79 | 78
  Day 3 | -1.1 [-6.0 to 3.8] | -11.3 [-16.2 to -6.4] | -10.2 [-15.2 to -5.2]
  Day 4: number analyzed (Participants) | 81 | 78 | 77
  Day 4 | -5.0 [-10.6 to 0.5] | -14.6 [-20.2 to -9.1] | -14.7 [-20.3 to -9.1]
  Day 5: number analyzed (Participants) | 72 | 82 | 81
  Day 5 | -9.5 [-15.8 to -3.2] | -16.1 [-22.3 to -9.9] | -17.6 [-23.9 to -11.3]
  Day 6: number analyzed (Participants) | 80 | 81 | 80
  Day 6 | -8.7 [-15.2 to -2.2] | -18.5 [-25.0 to -12.1] | -18.7 [-25.3 to -12.1]
  Day 7: number analyzed (Participants) | 79 | 81 | 80
  Day 7 | -12.3 [-19.4 to -5.2] | -20.0 [-27.1 to -12.9] | -18.8 [-26.0 to -11.6]
  Day 8: number analyzed (Participants) | 75 | 75 | 76
  Day 8 | -10.6 [-17.9 to -3.3] | -21.6 [-28.9 to -14.2] | -22.7 [-30.2 to -15.3]
  Day 9: number analyzed (Participants) | 83 | 75 | 80
  Day 9 | -9.9 [-17.6 to -2.3] | -20.9 [-28.7 to -13.2] | -21.7 [-29.5 to -13.9]
  Day 10: number analyzed (Participants) | 84 | 77 | 80
  Day 10 | -10.8 [-17.8 to -3.8] | -26.1 [-33.1 to -19.0] | -28.0 [-35.1 to -20.8]
  Day 11: number analyzed (Participants) | 79 | 77 | 74
  Day 11 | -10.7 [-17.7 to -3.7] | -26.5 [-33.5 to -19.4] | -26.3 [-33.5 to -19.1]
  Day 12: number analyzed (Participants) | 74 | 72 | 72
  Day 12 | -11.0 [-18.0 to -4.0] | -27.0 [-34.0 to -20.0] | -28.9 [-36.1 to -21.8]
  Day 13: number analyzed (Participants) | 80 | 80 | 77
  Day 13 | -14.1 [-20.4 to -7.8] | -25.2 [-31.5 to -18.8] | -32.5 [-39.0 to -26.0]
  Day 14: number analyzed (Participants) | 84 | 81 | 74
  Day 14 | -12.0 [-18.1 to -5.8] | -29.4 [-35.5 to -23.2] | -35.3 [-41.6 to -29.0]
  Day 15 | -15.8 [-22.7 to -8.8] | -30.7 [-37.7 to -23.7] | -33.4 [-40.5 to -26.3]

14. Secondary Outcome: Change From Baseline in Percentage Body Surface Area (BSA)
Description: BSA efficacy is derived from the sum of the BSA in handprints across 4 body regions assessed as part of the EASI assessment. Handprint refers to that of each individual participant for their own measurement. The BSA efficacy ranges from 0 to 100%, with higher values representing greater severity of AD. The percentage BSA ranges from 0 to 100, with higher scores representing greater severity of AD. Since the scalp, palms, and soles were excluded from the BSA (efficacy) assessment, the maximum possible percentage BSA was less than 100.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Units on a scale
  Week 2 | -10.9 [-14.0 to -7.8] | -21.0 [-24.1 to -17.9] | -20.7 [-23.8 to -17.6]
  Week 4 | -15.1 [-18.4 to -11.7] | -27.7 [-31.0 to -24.3] | -32.6 [-36.0 to -29.1]
  Week 8 | -21.8 [-25.3 to -18.3] | -32.6 [-36.1 to -29.1] | -34.1 [-37.7 to -30.6]
  Week 12 | -24.2 [-27.8 to -20.7] | -34.4 [-38.0 to -30.8] | -35.2 [-38.8 to -31.6]

15. Secondary Outcome: Percent Change From Baseline in Percentage BSA
Description: as for outcome 14
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Percent change
  Week 2 | -20.6 [-26.7 to -14.5] | -40.4 [-46.5 to -34.3] | -42.2 [-48.3 to -36.1]
  Week 4 | -29.0 [-36.3 to -21.8] | -55.4 [-62.7 to -48.1] | -66.0 [-73.4 to -58.6]
  Week 8 | -46.0 [-52.6 to -39.3] | -65.7 [-72.4 to -59.1] | -69.5 [-76.3 to -62.8]
  Week 12 | -53.4 [-60.1 to -46.7] | -71.4 [-78.2 to -64.7] | -72.6 [-79.3 to -65.8]

16. Secondary Outcome: Percentage of Participants Achieving Percentage BSA < 5% at Week 12
Description: as for outcome 14
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 94 | 89 | 93
Percentage of participants | 24.5 [15.8 to 33.2] | 38.2 [28.1 to 48.3] | 36.6 [26.8 to 46.3]

17. Secondary Outcome: Percentage of Participants Achieving Scoring Atopic Dermatitis (SCORAD) Response ≥ 50% Improvement From Baseline
Description: SCORAD is a validated scoring index for AD,which combines extent (0-100),severity (0-18),and subjective symptoms (0-20) based on pruritus and sleep loss,each scored (0-10). Extent,denoted as A,is measured by BSA affected by AD as a percentage of the whole BSA.The score for each body region is added up to determine A (maximum of 100).Severity, denoted as B,consists of the severity of several signs.Each is assessed as none(0),mild(1),moderate(2) or severe(3).The severity scores are added together to give B (maximum of 18).Subjective symptoms,denoted as C,are each scored by the participant using a NRS where "0" is no itch (or no sleeplessness) and "10" is the worst imaginable itch (or sleeplessness).These scores are added to give 'C' (maximum of 20).SCORAD for an individual is calculated by the formula: A/5 + 7B/2 + C (can range from 0 to 103).Higher values of SCORAD represent worse outcome.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 93 | 93
Percentage of participants
  Week 2: number analyzed (Participants) | 93 | 93 | 93
  Week 2 | 8.6 [2.9 to 14.3] | 22.6 [14.1 to 31.1] | 29.0 [19.8 to 38.3]
  Week 4: number analyzed (Participants) | 96 | 93 | 92
  Week 4 | 24.0 [15.4 to 32.5] | 44.1 [34.0 to 54.2] | 64.1 [54.3 to 73.9]
  Week 8: number analyzed (Participants) | 94 | 93 | 92
  Week 8 | 34.0 [24.5 to 43.6] | 65.6 [55.9 to 75.2] | 75.0 [66.2 to 83.8]
  Week 12: number analyzed (Participants) | 93 | 90 | 92
  Week 12 | 37.6 [27.8 to 47.5] | 75.6 [66.7 to 84.4] | 73.9 [64.9 to 82.9]

18. Secondary Outcome: Percentage of Participants Achieving SCORAD Response ≥ 75% Improvement From Baseline
Description: as for outcome 17
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 93 | 93
Percentage of participants
  Week 2: number analyzed (Participants) | 93 | 93 | 93
  Week 2 | 0 [0.0 to 3.9] | 5.4 [0.8 to 10.0] | 7.5 [2.2 to 12.9]
  Week 4: number analyzed (Participants) | 96 | 93 | 92
  Week 4 | 0 [0.0 to 3.8] | 11.8 [5.3 to 18.4] | 21.7 [13.3 to 30.2]
  Week 8: number analyzed (Participants) | 94 | 93 | 92
  Week 8 | 8.5 [2.9 to 14.2] | 17.2 [9.5 to 24.9] | 33.7 [24.0 to 43.4]
  Week 12: number analyzed (Participants) | 93 | 90 | 92
  Week 12 | 12.9 [6.1 to 19.7] | 36.7 [26.7 to 46.6] | 34.8 [25.1 to 44.5]

19. Secondary Outcome: Change From Baseline in SCORAD Total Score
Description: as for outcome 17
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 93
Units on a scale
  Week 2 | -12.3 [-15.4 to -9.2] | -24.6 [-27.7 to -21.6] | -25.8 [-28.9 to -22.7]
  Week 4 | -20.2 [-23.3 to -17.0] | -32.4 [-35.5 to -29.2] | -38.0 [-41.2 to -34.8]
  Week 8 | -26.6 [-30.0 to -23.2] | -37.3 [-40.7 to -33.9] | -41.5 [-45.0 to -38.0]
  Week 12 | -30.2 [-33.9 to -26.4] | -40.9 [-44.7 to -37.2] | -42.9 [-46.7 to -39.1]

20. Secondary Outcome: Percent Change From Baseline in SCORAD Total Score
Description: as for outcome 17
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 93
Percent change
  Week 2 | -18.7 [-23.1 to -14.2] | -36.1 [-40.6 to -31.7] | -38.7 [-43.2 to -34.2]
  Week 4 | -30.0 [-34.5 to -25.5] | -47.4 [-52.0 to -42.9] | -56.9 [-61.6 to -52.3]
  Week 8 | -39.9 [-44.9 to -34.8] | -54.0 [-59.0 to -48.9] | -62.0 [-67.2 to -56.9]
  Week 12 | -44.4 [-50.1 to -38.8] | -59.2 [-64.9 to -53.6] | -64.3 [-70.1 to -58.6]

21. Secondary Outcome: Change From Baseline in SCORAD Subjective Visual Analogue Scale (VAS) of Sleep Loss
Description: SCORAD is a validated scoring index for AD, which combines extent (A, 0-100), severity (B, 0-18), and subjective symptoms (C, 0-20) based on pruritus and sleep loss, each scored (0-10). The SCORAD for an individual is calculated by the formula: A/5 + 7B/2 + C (can range from 0 to 103). Subjective symptoms (ie, itch and sleep loss) are each scored by the participant using a VAS where "0" is no itch (or no sleep loss) and "10" is the worst imaginable itch (or sleep loss). The value for each should reflect the average on a 10 point scale for the last 3 days/nights. Changes from baseline in SCORAD subjective assessments of itch were not evaluated. Only changes from baseline in SCORAD subjective assessments of sleep loss are presented below.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 93
Units on a scale
  Week 2 | -0.9 [-1.4 to -0.4] | -2.1 [-2.6 to -1.6] | -2.6 [-3.1 to -2.1]
  Week 4 | -1.8 [-2.3 to -1.3] | -2.9 [-3.3 to -2.4] | -3.4 [-3.9 to -2.9]
  Week 8 | -2.2 [-2.7 to -1.7] | -3.3 [-3.8 to -2.9] | -3.7 [-4.2 to -3.2]
  Week 12 | -2.7 [-3.2 to -2.2] | -3.5 [-3.9 to -3.0] | -3.9 [-4.4 to -3.4]

22. Secondary Outcome: Percent Change From Baseline in SCORAD Subjective VAS of Sleep Loss
Description: as for outcome 21
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 93
Percent change
  Week 2 | 2.6 [-101.2 to 106.3] | 65.1 [-39.2 to 169.4] | -36.5 [-140.7 to 67.8]
  Week 4 | -20.0 [-35.2 to -4.9] | -35.2 [-50.7 to -19.8] | -53.4 [-69.1 to -37.8]
  Week 8 | -24.7 [-60.1 to 10.8] | -44.2 [-79.9 to -8.5] | -30.6 [-66.7 to 5.5]
  Week 12 | -39.5 [-77.7 to -1.3] | -49.8 [-88.3 to -11.3] | -35.2 [-74.1 to 3.7]

23. Secondary Outcome: Number of Days When a Corticosteroid Not Used up to Day 88
Time Frame: Baseline to Day 88
Population: The Full Analysis Set (FAS) included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. The analysis population included all participants in the FAS who had used corticosteroid during treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 83 | 89 | 82
Days | 6.8 [2.0 to 11.6] | 10.9 [6.2 to 15.5] | 15.1 [10.2 to 19.9]

24. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (DLQI)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items to assess participant-reported health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment).The DLQI is a psychometrically valid and reliable instrument that has been translated into several languages, and the DLQI total scores have been shown to be responsive to change. The minimally important difference for the DLQI has been estimated as a 3-5 point change from baseline. Each item is scored as "very much (3)", "a lot (2)", "a little (1)" and "not at all (0)". The score can range from 0 to 30. The higher values represent the worse dermatology life quality. Participants who withdrew from the study were counted as non-responder.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Units on a scale
  Week 2 | -4.2 [-5.1 to -3.3] | -6.1 [-7.1 to -5.2] | -6.3 [-7.2 to -5.3]
  Week 4 | -5.4 [-6.3 to -4.5] | -7.3 [-8.2 to -6.4] | -7.6 [-8.6 to -6.7]
  Week 8 | -6.1 [-7.0 to -5.1] | -8.1 [-9.1 to -7.1] | -8.2 [-9.2 to -7.2]
  Week 12 | -6.3 [-7.4 to -5.3] | -8.6 [-9.6 to -7.5] | -8.7 [-9.7 to -7.6]

25. Secondary Outcome: Percentage of Participants With ≥2.5 Points at Baseline and Achieving ≥2.5 Points Improvement From Baseline in Children's DLQI
Description: as for outcome 24
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 95 | 92 | 94
Percentage of participants
  Week 2: number analyzed (Participants) | 91 | 91 | 94
  Week 2 | 61.5 [51.5 to 71.5] | 73.6 [64.6 to 82.7] | 71.3 [62.1 to 80.4]
  Week 4: number analyzed (Participants) | 95 | 91 | 94
  Week 4 | 73.7 [64.8 to 82.5] | 82.4 [74.6 to 90.2] | 73.4 [64.5 to 82.3]
  Week 8: number analyzed (Participants) | 93 | 92 | 93
  Week 8 | 71.0 [61.7 to 80.2] | 85.9 [78.8 to 93.0] | 79.6 [71.4 to 87.8]
  Week 12: number analyzed (Participants) | 93 | 89 | 93
  Week 12 | 67.7 [58.2 to 77.2] | 80.9 [72.7 to 89.1] | 78.5 [70.1 to 86.8]

26. Secondary Outcome: Change From Baseline in Anxiety of Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a 14-item patient reported outcome (PRO) measure used to detect states of anxiety and depression over the past week. Seven of the items relate to anxiety and seven relate to depression. Each item is scored from 0 to 3 which means a person can score between 0 to 21 for either anxiety or depression. Higher values represent worse outcome.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Units on a scale
  Week 2 | -1.2 [-1.7 to -0.7] | -1.6 [-2.1 to -1.1] | -1.3 [-1.8 to -0.8]
  Week 4 | -1.5 [-2.1 to -1.0] | -1.6 [-2.2 to -1.1] | -1.9 [-2.5 to -1.3]
  Week 8 | -1.7 [-2.3 to -1.1] | -2.1 [-2.7 to -1.5] | -2.2 [-2.8 to -1.5]
  Week 12 | -2.1 [-2.7 to -1.5] | -2.0 [-2.6 to -1.4] | -2.4 [-3.0 to -1.8]

27. Secondary Outcome: Change From Baseline in Depression of HADS
Description: as for outcome 26
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Units on a scale
  Week 2 | -0.8 [-1.3 to -0.3] | -1.2 [-1.7 to -0.8] | -0.8 [-1.3 to -0.3]
  Week 4 | -0.8 [-1.3 to -0.3] | -1.3 [-1.8 to -0.8] | -1.3 [-1.8 to -0.8]
  Week 8 | -1.1 [-1.6 to -0.6] | -1.4 [-1.9 to -0.9] | -1.2 [-1.7 to -0.7]
  Week 12 | -1.0 [-1.5 to -0.5] | -1.4 [-1.9 to -0.8] | -1.2 [-1.7 to -0.6]

28. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM)
Description: The POEM is a 7-item PRO measure used to assess the impact of AD over the past week. Each item is scored as "no days (0)", "1-2 days (1)", "3-4 days (2)", "5-6 days (3)" and "every day (4)". The score ranges from 0 to 28. The higher values represent more severe AD.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Placebo: Participants received PF-04965842-matching placebo tablets QD
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 95 | 95 | 94
Units on a scale
  Week 2 | -3.4 [-4.7 to -2.1] | -6.9 [-8.2 to -5.6] | -8.2 [-9.5 to -6.9]
  Week 4 | -4.8 [-6.0 to -3.6] | -9.5 [-10.7 to -8.3] | -10.6 [-11.9 to -9.4]
  Week 8 | -5.4 [-6.7 to -4.0] | -10.0 [-11.4 to -8.7] | -10.6 [-12.0 to -9.3]
  Week 12 | -6.9 [-8.3 to -5.6] | -11.1 [-12.5 to -9.7] | -10.9 [-12.2 to -9.5]

29. Secondary Outcome: Change From Baseline in Dermatitis Family Impact (DFI) at Week 12
Description: The DFI is a validated 10-item measure filled out by the parent/caregiver of the patient used to assess the impact of the patient's eczema on the family. The instrument has a recall period of 7 days. Each item is scored as "very much (3)", "a lot (2)", "a little (1)" or "not at all (0)". The score can range from 0 to 30. The higher values represent the worse impact.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 92 | 95 | 93
Units on a scale | -5.2 [-6.5 to -3.9] | -6.7 [-7.9 to -5.4] | -7.3 [-8.6 to -6.0]

30. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA)
Description: The PtGA asked the participant to evaluate the overall cutaneous disease at that point in time on a single-item, 5-point scale. The same category labels used in the IGA were used for the PtGA, ie, "severe (4)", "moderate (3)", "mild (2)","almost clear (1)", and "clear (0)". The PtGA was completed as per schedule of activities.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Units on a scale
  Week 2 | -0.4 [-0.6 to -0.3] | -0.7 [-0.9 to -0.6] | -1.0 [-1.1 to -0.8]
  Week 4 | -0.7 [-0.8 to -0.5] | -0.9 [-1.1 to -0.8] | -1.2 [-1.4 to -1.1]
  Week 8 | -0.8 [-1.0 to -0.6] | -1.2 [-1.3 to -1.0] | -1.4 [-1.6 to -1.2]
  Week 12 | -0.9 [-1.1 to -0.7] | -1.4 [-1.6 to -1.2] | -1.6 [-1.8 to -1.4]

31. Secondary Outcome: Percentage of Participants With ≥2 Points at Baseline and Achieving 'Clear' or 'Almost Clear' and ≥2 Points Improvement From Baseline in PtGA
Description: as for outcome 30
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number of Participants Analyzed refers to the number of participants evaluable for this outcome measure. Number analyzed refers to the number of participants evaluable for each time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 93 | 94
Percentage of participants
  Week 2: number analyzed (Participants) | 92 | 92 | 94
  Week 2 | 1.1 [0.0 to 3.2] | 5.4 [0.8 to 10.1] | 5.3 [0.8 to 9.9]
  Week 4: number analyzed (Participants) | 96 | 92 | 94
  Week 4 | 4.2 [0.2 to 8.2] | 14.1 [7.0 to 21.2] | 20.2 [12.1 to 28.3]
  Week 8: number analyzed (Participants) | 94 | 93 | 93
  Week 8 | 6.4 [1.4 to 11.3] | 22.6 [14.1 to 31.1] | 26.9 [17.9 to 35.9]
  Week 12: number analyzed (Participants) | 94 | 90 | 93
  Week 12 | 10.6 [4.4 to 16.9] | 30.0 [20.5 to 39.5] | 36.6 [26.8 to 46.3]

32. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension Youth Scale (EQ-5D-Y) VAS Score
Description: The EQ-5D is a validated, standardized, generic instrument that is the most widely used preference based health related quality of life questionnaire in cost effectiveness and health technologies assessment. The EQ-5D-Y is a version of the instrument specifically developed and validated for use by youths aged 12 through 17 years. Components assess level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety and depression. Score scale for each domain ranges from 1 (minimum) to 3 (maximum), with higher scores indicating worse health condition. In addition, respondents use a vertical, graduated Visual Analogue Scale (VAS) to rate their own health between 0 (the worst) and 100 (the best health state he/she can imagine).
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Units on a scale
  Week 2 | 7.140 [3.787 to 10.492] | 11.241 [7.882 to 14.601] | 12.141 [8.763 to 15.520]
  Week 4 | 8.784 [5.625 to 11.943] | 13.222 [10.020 to 16.423] | 14.677 [11.438 to 17.917]
  Week 8 | 8.415 [4.888 to 11.941] | 14.502 [10.977 to 18.028] | 14.653 [11.076 to 18.231]
  Week 12 | 9.944 [6.373 to 13.515] | 14.226 [10.624 to 17.828] | 15.756 [12.153 to 19.360]

33. Secondary Outcome: Change From Baseline in Pediatric Functional Assessment of Chronic Illness Therapy Fatigue Scale (Peds-FACIT-F) at Week 12
Description: The Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-F) is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (none of the time) to 4 (all of the time). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-F score for a total possible score of 0 (worse score) to 52 (better score), with higher scores representing better overall health status (less fatigue). Changes from baseline at Week 12 are presented below. Changes from baseline at other scheduled time points were not evaluated.
Time Frame: Baseline to Week 12
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Units on a scale | 2.5 [1.1 to 3.9] | 4.5 [3.0 to 5.9] | 4.3 [2.9 to 5.7]

34. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. TEAEs were AEs that occurred following the start of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator.
Time Frame: 16 weeks
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Participants
  All-causality TEAEs | 50 | 54 | 59
  Treatment-related TEAEs | 16 | 20 | 31

35. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. Treatment-related SAEs were determined by the investigator.
Time Frame: 16 weeks
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Participants
  All-causality SAEs | 2 | 0 | 1
  Treatment-related SAEs | 0 | 0 | 0

36. Secondary Outcome: Number of Participants Who Discontinued From the Study Due to TEAEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. TEAEs were AEs that occurred following the start of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator.
Time Frame: 16 weeks
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 94
Participants
  All-causality TEAEs | 2 | 1 | 2
  Treatment-related TEAEs | 0 | 0 | 2

37. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory tests included hematology (including coagulation panel), clinical chemistry, lipid profile panel, and routine urinalysis. LLN is lower limit of normal. ULN is upper limit of normal.
Time Frame: 16 weeks
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number of Participants Analyzed refers to the number of participants who were evaluable for this outcome measure. Number analyzed refers to the number of participants with at least one observation of the given laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 93
Participants
  Hemoglobin (g/dL) <0.8*LLN | 0 | 0 | 0
  Hematocrit (%) <0.8*LLN: number analyzed (Participants) | 96 | 93 | 93
  Hematocrit (%) <0.8*LLN | 0 | 0 | 0
  Erythrocytes (10^6/mm^3) <0.8*LLN | 0 | 0 | 0
  Reticulocytes (10^3/mm^3) <0.5*LLN: number analyzed (Participants) | 68 | 68 | 70
  Reticulocytes (10^3/mm^3) <0.5*LLN | 0 | 0 | 0
  Reticulocytes (10^3/mm^3) >1.5*ULN: number analyzed (Participants) | 68 | 68 | 70
  Reticulocytes (10^3/mm^3) >1.5*ULN | 0 | 0 | 0
  Ery. Mean Corpuscular Volume (10^-15L) <0.9*LLN: number analyzed (Participants) | 96 | 93 | 93
  Ery. Mean Corpuscular Volume (10^-15L) <0.9*LLN | 1 | 1 | 0
  Ery. Mean Corpuscular Volume (10^-15L) >1.1*ULN: number analyzed (Participants) | 96 | 93 | 93
  Ery. Mean Corpuscular Volume (10^-15L) >1.1*ULN | 0 | 0 | 0
  Ery. Mean Corpuscular Hemoglobin (pg/cell) <0.9*LLN | 1 | 1 | 0
  Ery. Mean Corpuscular Hemoglobin (pg/cell) >1.1*ULN | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration (g/dL) <0.9*LLN: number analyzed (Participants) | 96 | 93 | 93
  Ery. Mean Corpuscular HGB Concentration (g/dL) <0.9*LLN | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration (g/dL) >1.1*ULN: number analyzed (Participants) | 96 | 93 | 93
  Ery. Mean Corpuscular HGB Concentration (g/dL) >1.1*ULN | 0 | 0 | 0
  Platelets (10^3/mm^3) <0.5*LLN | 1 | 0 | 0
  Platelets (10^3/mm^3) >1.75*ULN | 0 | 0 | 0
  Reticulocytes/Erythrocytes (%) <0.5*LLN: number analyzed (Participants) | 68 | 68 | 70
  Reticulocytes/Erythrocytes (%) <0.5*LLN | 0 | 0 | 0
  Reticulocytes/Erythrocytes (%) >1.5*ULN: number analyzed (Participants) | 68 | 68 | 70
  Reticulocytes/Erythrocytes (%) >1.5*ULN | 0 | 0 | 1
  Leukocytes (10^3/mm^3) <0.6*LLN | 0 | 0 | 0
  Leukocytes (10^3/mm^3) >1.5*ULN | 1 | 0 | 0
  Lymphocytes (10^3/mm^3) <0.8*LLN | 0 | 0 | 1
  Lymphocytes (10^3/mm^3) >1.2*ULN | 0 | 0 | 1
  Lymphocytes/Leukocytes (%) <0.8*LLN | 6 | 4 | 6
  Lymphocytes/Leukocytes (%) >1.2*ULN | 1 | 1 | 4
  Neutrophils (10^3/mm^3) <0.8*LLN | 1 | 2 | 1
  Neutrophils (10^3/mm^3) >1.2*ULN | 6 | 5 | 3
  Neutrophils/Leukocytes (%) <0.8*LLN | 5 | 3 | 7
  Neutrophils/Leukocytes (%) >1.2*ULN | 0 | 0 | 0
  Basophils (10^3/mm^3) >1.2*ULN | 3 | 0 | 0
  Basophils/Leukocytes (%) >1.2*ULN | 35 | 24 | 27
  Eosinophils (10^3/mm^3) >1.2*ULN | 63 | 55 | 39
  Eosinophils/Leukocytes (%) >1.2*ULN | 61 | 62 | 47
  Monocytes (10^3/mm^3) >1.2*ULN | 1 | 0 | 0
  Monocytes/Leukocytes (%) >1.2*ULN | 7 | 11 | 6
  Activated Partial Thromboplastin Time (sec) >1.1*ULN | 2 | 4 | 4
  Prothrombin Time (sec) >1.1*ULN | 4 | 6 | 8
  Prothrombin Intl.Normalized Ratio >1.1*ULN | 0 | 0 | 0
  Bilirubin (mg/dL) >1.5*ULN | 1 | 4 | 0
  Direct Bilirubin (mg/dL) >1.5*ULN: number analyzed (Participants) | 96 | 93 | 93
  Direct Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 0
  Indirect Bilirubin (mg/dL) >1.5*ULN: number analyzed (Participants) | 96 | 93 | 93
  Indirect Bilirubin (mg/dL) >1.5*ULN | 1 | 2 | 0
  Aspartate Aminotransferase (U/L) >3.0*ULN | 1 | 1 | 3
  Alanine Aminotransferase (U/L) >3.0*ULN | 0 | 3 | 1
  Gamma Glutamyl Transferase (U/L) >3.0*ULN | 1 | 0 | 0
  Lactate Dehydrogenase (U/L) >3.0*ULN | 0 | 1 | 2
  Alkaline Phosphatase (U/L) >3.0*ULN | 0 | 0 | 1
  Protein (g/dL) <0.8*LLN | 0 | 0 | 0
  Protein (g/dL) >1.2*ULN | 0 | 0 | 1
  Albumin (g/dL) <0.8*LLN | 0 | 0 | 0
  Albumin (g/dL) >1.2*ULN | 0 | 0 | 3
  Urea Nitrogen (mg/dL) >1.3*ULN | 0 | 0 | 0
  Creatinine (mg/dL) >1.3*ULN | 3 | 2 | 0
  Urate (mg/dL) >1.2*ULN | 2 | 4 | 1
  LDL Cholesterol (mg/dL) >1.2*ULN | 2 | 2 | 3
  Triglycerides (mg/dL) >1.3*ULN | 17 | 11 | 13
  Sodium (mEq/L) <0.95*LLN | 0 | 0 | 0
  Sodium (mEq/L) >1.05*ULN | 0 | 0 | 0
  Potassium (mEq/L) <0.9*LLN | 0 | 0 | 0
  Potassium (mEq/L) >1.1*ULN | 1 | 0 | 0
  Chloride (mEq/L) <0.9*LLN | 0 | 0 | 0
  Chloride (mEq/L) >1.1*ULN | 0 | 0 | 0
  Calcium (mg/dL) <0.9*LLN | 0 | 0 | 0
  Calcium (mg/dL) >1.1*ULN | 0 | 0 | 0
  Bicarbonate (mEq/L) <0.9*LLN | 1 | 1 | 0
  Bicarbonate (mEq/L) >1.1*ULN | 0 | 0 | 0
  Glucose (mg/dL) <0.6*LLN | 0 | 0 | 0
  Glucose (mg/dL) >1.5*ULN | 0 | 2 | 3
  Creatine Kinase (U/L) >2.0*ULN | 5 | 7 | 12
  Cholesterol (mg/dL)>1.3*ULN | 2 | 2 | 2
  HDL Cholesterol (mg/dL) <0.8*LLN | 0 | 0 | 0
  Urine Specific Gravity (scalar) <1.003: number analyzed (Participants) | 0 | 1 | 2
  Urine Specific Gravity (scalar) <1.003 | 0 | 0 | 0
  Urine Specific Gravity (scalar) >1.030: number analyzed (Participants) | 0 | 1 | 2
  Urine Specific Gravity (scalar) >1.030 | 0 | 1 | 0
  Urine pH (Scalar) <4.5 | 0 | 0 | 0
  Urine pH (Scalar) >8 | 0 | 1 | 0
  Urine Glucose >=1 | 1 | 0 | 0
  Urine Ketones >=1 | 8 | 0 | 1
  Urine Protein >=1 | 4 | 5 | 0
  Urine Hemoglobin >=1 | 20 | 19 | 15
  Urine Nitrite >=1 | 0 | 1 | 0
  Urine Leukocyte Esterase >=1 | 7 | 14 | 17
  Urine Erythrocytes (/HPF) >=20: number analyzed (Participants) | 49 | 41 | 44
  Urine Erythrocytes (/HPF) >=20 | 8 | 7 | 5
  Urine Leukocytes (/HPF) >=20: number analyzed (Participants) | 57 | 62 | 54
  Urine Leukocytes (/HPF) >=20 | 0 | 2 | 1
  Urine Granular Casts (/LPF) >1: number analyzed (Participants) | 1 | 0 | 0
  Urine Granular Casts (/LPF) >1 | 1 | 0 | 0
  Urine Hyaline Casts (/LPF) >1: number analyzed (Participants) | 4 | 3 | 3
  Urine Hyaline Casts (/LPF) >1 | 2 | 1 | 1
  Urine Bacteria >20: number analyzed (Participants) | 18 | 22 | 18
  Urine Bacteria >20 | 0 | 0 | 0

38. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Prespecified Criteria
Description: A 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT intervals. All scheduled ECGs were performed after the participant had rested quietly for at least 10 minutes in a supine position. Reading of ECGs were performed by a central reader who has expertise reading and interpreting ECGs in adolescents. The QTcF interval is the only prespecified ECG criteria (Marked prolongation of the QTcF interval to >500 ms or >60 ms change from screening ECG); data are presented below.
Time Frame: 16 weeks
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Number of Participants Analyzed refers to the number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 93
Participants
  QTcF Interval, Single Beat (msec) Value >500 | 0 | 0 | 0
  QTcF Interval, Single Beat (msec) Change From Screening >60 | 0 | 0 | 0

39. Secondary Outcome: Categorization of Vital Signs Data Meeting Prespecified Criteria
Description: Vital signs (pulse rate, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes.
Time Frame: 16 weeks
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 96 | 95 | 93
Participants
  Diastolic Blood Pressure Value <50mmHg | 3 | 1 | 9
  Diastolic Blood Pressure Increase From Baseline >= 20mmHg | 3 | 6 | 6
  Diastolic Blood Pressure Decrease From Baseline >= 20mmHg | 3 | 4 | 8
  Pulse Rate Value <40 bpm | 0 | 0 | 0
  Pulse Rate Value >120 bpm | 0 | 0 | 0
  Systolic Blood Pressure Value <90mmHg | 4 | 7 | 4
  Systolic Blood Pressure Increase From Baseline >=30mmHg | 2 | 1 | 2
  Systolic Blood Pressure Decrease From Baseline >=30mmHg | 2 | 1 | 2

40. Secondary Outcome: Fold Increase of Immunoglobulin G (IgG) Concentrations Against Specific Vaccine Antigens at 4 Weeks Post-Vaccination
Description: The immunogenicity analysis was to evaluate the effect of abrocitinib on immunogenicity to a tetanus, diphtheria and pertussis combination vaccine (Tdap) vaccine in adolescent participants 12 to <18 years of age with moderate to severe AD. Participants who completed 8 weeks of treatment with study intervention received Tdap at Week 8, and had blood samples collected for the evaluation of immunogenicity to the vaccine at Weeks 8 and 12. The fold increase was defined as the ratio (post-vaccination: pre-vaccination) of concentration values. The geometric mean fold rise (GMFR) is presented below, and was calculated by first arithmetically averaging the logarithmically transformed ratio (post-vaccination: pre-vaccination) values, and then back transformation. A 95% CI for GMFR was constructed by back transformation of the CI for the logarithmically transformed GMFRs computed using the Student's t distribution.
Time Frame: 4 weeks post-vaccination with Tdap (Week 12)
Population: The immunogenicity sub-study analysis set included all participants who had completed 8 weeks of treatment and received Tdap vaccination. Number of Participants Analyzed refers to the number of participants evaluable in the analysis set at the specified visit.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 10 | 8 | 4
Ratio
  Diphtheria IgG Antibody | 14.00 [6.32 to 30.99] | 6.51 [2.31 to 18.34] | 34.61 [6.96 to 172.06]
  Filamentous Hemagglutinin IgG | 15.19 [4.89 to 47.16] | 11.48 [2.65 to 49.69] | 22.77 [7.26 to 71.45]
  Fimbriae 2/3 IgG | 1.93 [0.79 to 4.73] | 1.11 [0.85 to 1.46] | 1.47 [0.61 to 3.50]
  Pertactin IgG | 54.03 [14.67 to 199.03] | 15.60 [5.77 to 42.14] | 60.18 [12.79 to 283.08]
  Pertussis Toxin IgG | 6.94 [1.95 to 24.71] | 10.17 [4.71 to 21.94] | 33.16 [5.04 to 218.38]
  Tetanus Toxoid IGG AB | 8.36 [1.62 to 43.18] | 16.26 [3.52 to 75.11] | 48.41 [9.01 to 260.09]

41. Secondary Outcome: Plasma PF-04965842 Concentration at Week 8
Time Frame: 2 hours pre-dose at Week 8
Population: The PK analysis included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Samples from site 1173 were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 72 | 62
ng/mL | 7.882 (26.350) | 32.33 (76.506)

42. Secondary Outcome: Plasma PF-04965842 Concentration at Week 12
Time Frame: 2 hours post-dose at Week 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 59 | 50
ng/mL | 486.6 (403.69) | 1271 (1000.4)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Placebo | PF-04965842 100mg QD | PF-04965842 200mg QD
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/95 | 0/94
Serious Adverse Events (participants affected / at risk) | 2/96 | 0/95 | 1/94
Other Adverse Events (participants affected / at risk) | 42/96 | 40/95 | 50/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=96) | PF-04965842 100mg QD (N=95) | PF-04965842 200mg QD (N=94)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis stopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=96) | PF-04965842 100mg QD (N=95) | PF-04965842 200mg QD (N=94)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 7 (7) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 4 (5) | 4 (4)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 6 (9)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 5 (5)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (6) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 5 (7) | 8 (12)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood uric acid increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Protein urine (Investigations) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (11) | 8 (10) | 8 (9)
Oral herpes (Infections and infestations) | 0 (0) | 1 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (3) | 5 (5) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 10 (12) | 9 (11) | 10 (14)
Pyrexia (General disorders) | 4 (4) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 7 (7) | 17 (27)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT03796676/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT03796676/SAP_001.pdf